CLINICAL TRIAL: NCT04620746
Title: Validate an Easy to Administer Algorithm to Define Penicillin (PCN-B-lactam) Allergy Status in Sexually Transmitted Disease (STD) Clinic Outpatients
Brief Title: Penicillin Allergy Testing in STD Clinics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Indiana University School of Medicine (Other); Wake Forest University Health Sciences (Other); Louisiana State University Health Sciences Center in New Orleans (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00220384; HHSN272201300012I/HHSN27200015 (Other Grant/Funding Number: National Institute Of Allergy & Infectious Disease)
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Penicillin Allergy
MeSH Terms: interventions — Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Skin Testing Arm (Active Comparator): These subjects with reported PCN allergy and reported low risk responses will receive skin testing followed by oral challenge
  Interventions: Drug: Penicillin Major Determinant (PrePen) Skin Testing; Drug: Direct Oral challenge
- Direct Oral Challenge (Active Comparator): These subjects with reported PCN allergy and low risk responses will bypass skin testing and have direct oral challenge with amoxicillin
  Interventions: Drug: Direct Oral challenge

INTERVENTIONS:
Drug: Penicillin Major Determinant (PrePen) Skin Testing — Skin testing followed by oral challenge with amoxicillin 250 mg single dose
  Other Names: Penicillin G Minor Determinant Skin Testing
  Arms: Skin Testing Arm
Drug: Direct Oral challenge — Direct oral challenge with test dose of amoxicillin 25mg followed by amoxicillin 250mg single dose

SUMMARY:
Demonstration project to implement penicillin allergy testing in STD outpatients using a questionnaire and pen allergy testing

DETAILED DESCRIPTION:
all subjects receive risk questionnaire For subjects without high risk responses, randomized to direct oral challenge or PCN skin testing followed by oral challenge

ELIGIBILITY:
Inclusion Criteria:

* Prior history of PCN allergy

Exclusion Criteria:

* No immunodeficiency or contraindication to skin testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Zenilman, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Louisiana State University, New Orleans, Louisiana
  - University of Washington-Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Blinded data set is available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be uploaded and provided when study is completed and analyzed. Completed May 2023

REFERENCES:
- [Derived] Lillis RA, Barbee LA, McNeil CJ, Newman L, Fortenberry JD, Alvarez-Arango S, Zenilman JM. Randomized Multicenter Trial for the Validation of an Easy-to-Administer Algorithm to Define Penicillin Allergy Status in Sexually Transmitted Infection Clinic Outpatients. Clin Infect Dis. 2024 May 15;78(5):1131-1139. doi: 10.1093/cid/ciae064. PMID 38325290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 4 STI clinics. Enrollment criteria were whether they reported a history of having had, or been told that they have penicillin or beta-lactam allergy
Pre-assignment Details: All participants were administered a risk questionnaire to determine whehter they were classfied as high-risk or low risk for true penicillin allergy, based on input from allergy experts. Subjects who ahd a high risk history (eg hives within past 5 years) were referred for further allergist evaluation, as they were deemed too high risk to be evaluated further in an STI clinic
Period: Overall Study
Arm/Group | Skin Testing Arm | Direct Oral Challenge
Started | 139 | 145
Completed | 136 | 144
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Uniterpretable skin test | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Skin Testing Arm | Direct Oral Challenge | Total
Number analyzed (Participants) | 139 | 145 | 284
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 137 | 143 | 280
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 35.9 [19 to 68] | 37.4 [18 to 67] | 36.6 [18 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 41 | 86
  Male | 94 | 104 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 15 | 34
  Not Hispanic or Latino | 117 | 130 | 247
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 9
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 29 | 42 | 71
  White | 104 | 90 | 194
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 139 | 145 | 284

OUTCOME MEASURES:

1. Primary Outcome: Number of Respondents Who Responded YES to Any Question Defining High Risk Penicillin Allergy Using Questionnaire Developed by the Study
Description: Used yes/no questionnaire designed by study team. Any positive response on the high-risk history was grounds for exclusion from randomization to allergy testing arm
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Skin Testing Arm: These subjects with reported PCN allergy and reported low risk responses will receive skin testing followed by oral challenge
  Penicillin Major Determinant (PrePen) Skin Testing: Skin testing followed by oral challenge with amoxicillin 250 mg single dose
  Direct Oral challenge: Direct oral challenge with amoxicillin 250mg single dose
Arm/Group | Skin Testing Arm | Direct Oral Challenge
Number analyzed (Participants) | 139 | 145
Participants | 36 | 36

2. Primary Outcome: Safety of Direct Oral Challenge Defined by Number of Subjects Who Did Not Have Pre-defined Changes in Vital Signs or Pre-defined Emergence of New Respiratory or Skin Symptoms After Oral Challenge
Description: Safety was determined by the presence or absence of adverse reactions. Symptoms assessed included pruritis, flushing, shortness of breath. Physical examination included vital signs, blood pressure, pulse, respiratory rate and peak expiratory flow
Time Frame: 30 minutes after intervention
Population: Number of participants analyzed is the number who completed the testing modalities
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Testing Arm | Direct Oral Challenge
Number analyzed (Participants) | 99 | 103
Participants | 96 | 95
Statistical Analysis 1: Comparison: Skin Testing Arm vs Direct Oral Challenge; Test type: Superiority; p = 0.98, Chi-squared, Corrected

3. Secondary Outcome: Patient Acceptability of PCN Testing/Oral Challenge Assessed by a Study Team Developed Questionnaire
Description: Brief Acceptabilty Questionnaire to subjects on acceptability of PCN allergy testing in the STD clinic setting. Reported as number of participants who found testing acceptable. Questionnaire asked subjects whether they found the process helpful and whether they would return for this type of testing. Using a 1-5 scale, with 1 defined as extremely helpful and 5 defined as not helpful.
Time Frame: Immediately after intervention
Population: The numbers reflected in Participants Analyzed for this outcome represent the number of participants who completed the Acceptability questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- Skin Testing Arm: Skin testing followed by oral challenge with amoxicillin 250 mg single dose
  Direct Oral challenge: Direct oral challenge with test dose of amoxicillin 25mg followed by amoxicillin 250mg single dose
Arm/Group | Skin Testing Arm | Direct Oral Challenge
Number analyzed (Participants) | 99 | 89
Participants | 99 | 89
Statistical Analysis 1: Comparison: Skin Testing Arm vs Direct Oral Challenge; Test type: Superiority; p = 0.95, Chi-squared

4. Secondary Outcome: Provider Assessment of Feasibility of Allergy Evaluation at the End of Study
Description: Provider assessment of feasibility of providing PCN testing in the STD clinic setting. This was based on a team-developed questionnaire using Likert scale questions that asked about feasibility and self-efficacy in performing the assessments. Feasibility defined by 1-5 scale, with 1= highly feasible and 5=not feasible. Reported as number of providers who found PCN testing feasible.
Time Frame: 18 months
Population: Response to questionnaire was optional
Measure: Count of Participants; unit: Participants
Groups:
- Providers: Providers who paricpated in the study
Arm/Group | Providers
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse events were recorded up to 1 week post intervention
Arm/Group | Skin Testing Arm | Direct Oral Challenge
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/145
Other Adverse Events (participants affected / at risk) | 16/139 | 13/145
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skin Testing Arm (N=139) | Direct Oral Challenge (N=145)
Minor adverse events (Immune system disorders) | 16 (16) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT04620746/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT04620746/SAP_001.pdf
  • Informed Consent Form (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT04620746/ICF_002.pdf